CLINICAL TRIAL: NCT07306039
Title: Feasibility of eLi12 in a Clinical Setting
Brief Title: Feasibility of eLi12
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ole Köhler-Forsberg (Other)
Collaborators: Randers Regional Hospital (Other); Gødstrup Hospital (Other)
Responsible Party: Sponsor-Investigator, Ole Köhler-Forsberg, MD, PhD, Associate Professor, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025_eLi12
Record Dates: First submitted 2025-12-03; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder (BD)
Keywords: Lithium; Trough level; Clinical feasibility; eLi12
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to have shown eLi12 (the estimated 12-hour lithium blood concentration) or not. All participants will have shown usual lithium concentration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants will have shown eLi12 (Active Comparator): Participants and their treating clinicians will have shown eLi12, the estimated 12-hour lithium concentration, in the electronic patient journal on top of the usual Se-Li concentration
  Interventions: Procedure: Participants will have shown eLi12
- Participants will not have shown eLi12 (Placebo Comparator): Participants will not have shown eLi12, the estimated 12-hour lithium concentration, in the electronic patient journal but only the usual Se-Li concentration
  Interventions: Procedure: Participants will not have shown eLi12

INTERVENTIONS:
Procedure: Participants will have shown eLi12 — Participants will have shown eLi12, the estimated 12-hour lithium level, in the electronic patient journal
  Arms: Participants will have shown eLi12
Procedure: Participants will not have shown eLi12 — Participants will not have shown eLi12, the estimated 12-hour lithium level, in the electronic patient journal
  Arms: Participants will not have shown eLi12

SUMMARY:
eLi12 represents a new method to estimate the serum-lithium (Se-Li) concentration at 12 hours after the most recent lithium dose. eLi12 is a mathematical equation that presents the clinician with an estimated 12-hour Se-Li level when the lithium blood test is not taken 12 hours after the most recent lithium dose, but e.g., after 8 or 16 hours. The eLi12 equation is based on a development study and supported by two independent proof-of-concept studies. In these studies, eLi12 estimated a Se-Li concentration that was significantly closer to the 12-hour Se-Li level compared to the actual measured Se-Li in all scenarios between 3 hours and 24 hours after the most recent lithium dose. Before eLi12 can be implemented into a clinical setting, it needs to be tested whether lithium-treated patients actually can register the time for the last lithium intake (prerequisite for eLi12) and if eLi12 can provide improvements for everyday clinical work. The objective of this study is to test 1) whether lithium-treated patients can register the time of the most recent lithium intake at the time of their lithium blood test (which is a necessary data point for the eLi12 equation), 2) the difference between eLi12 and Se-Li, 3) if eLi12 will have less variation compared to the actual measured Se-Li concentrations, 4) patient satisfaction with the eLi12 solution and self-reported symptoms, and 5) clinician satisfaction with the eLi12 solution.

DETAILED DESCRIPTION:
Hypothesis The main hypotheses are that 1) the majority (>80%) of patients will register the time since the last lithium dose, 2) there will be a difference between eLi12 and Se-Li among participants who got the lithium blood test at a different time point than 12 hours after the last dose, 3) eLi12 will show less variation compared to the measured lithium concentration, 4) patients will be satisfied with a solution that gives more flexibility regarding blood test timing and will have slightly fewer self-reported symptoms and better quality of life, and 5) clinicians will be satisfied with the eLi12 solution.

Study design Quality assurance study testing the feasibility of eLi12. Patients Patients with a bipolar disorder diagnosis (ICD-10: F30-31) treated with lithium (ATC-code: N05AN01) aged ≥18 years and followed at the bipolar disorder outpatient clinic at AUHP, the outpatient clinic for affective disorders at Randers Psychiatric Hospital, or the outpatient clinic for affective disorders at Gødstrup Psychiatric Hospital.

Procedures The lithium treatment and all blood tests are based on clinical indication prescribed by a clinician independent of the present study with the time for the blood test being booked by the patient (i.e., all independent of the present study protocol representing real-world clinical practice). eLi12 is a new method to estimate the 12-hour Se-Li level when the lithium blood test is not taken 12 hours after the most recent lithium dose. Implementation of eLi12 requires that lithium-treated patients register the time for the most recent lithium intake (i.e., the time when they took their last lithium dose the evening before the blood test) at the time of their lithium blood test. Using the already available data on 1) the Se-Li concentration measured at 2) the time-point of the blood test, the patient-reported time since the last lithium dose can then be used to calculate the eLi12 value. Participants in the present study will be randomized to have their eLi12 value presented in the electronic patient journal MidtEPJ. This means that the measured Se-Li will always be presented (i.e., standard clinical practice will continue as usual), and for 50% of participants, the eLi12 value will also be presented. Hence, during participation in this study, patients will be randomized to either have eLi12 shown together with their usual Se-Li measurement or to only have the Se-Li measurement presented (i.e., treatment-as-usual without the eLi12 estimation). This means that all participants will follow treatment-as-usual with 50% receiving additional information via eLi12. The present study will investigate the feasibility of eLi12 implementation and acquire new data about eLi12, but not acquire new knowledge about lithium as a drug.

Follow-up The study will be conducted from Q4 2025 until December 31, 2027. Individual participation will occur from the date of inclusion until the end of the study. The proposed study period is deemed necessary in order to ensure sufficient time for recruitment and to ensure several blood tests from the same individual to allow for testing the individual variation in Se-Li and eLi12. Patients will be treated and followed according to normal clinical treatment guidelines at the clinic. It will always be up to the attending clinician to evaluate whether a new dose (i.e., increase or decrease of the present lithium dose) is necessary and relevant.

Endpoints The study will evaluate three co-primary outcomes: 1) The percentage of patients registering the time since the last lithium dose, 2) the difference between eLi12 and Se-Li, and 3) for those periods of time where participants have no change in their lithium dose, the variation in eLi12 compared to the actual measured lithium concentrations at ≤10 hours or ≥14 hours from the last dose.

Secondary outcome measures will include 1) questionnaires filled out before and after participation in the study by the participants whether they prefer a solution as eLi12 that gives more flexibility with regards to timing of lithium blood tests, 2) questionnaires filled out regularly by the attending clinicians reporting whether eLi12 is a safe and intuitive solution, and 3) changes on questionnaires filled out by participants before and after the study measuring self-reported symptoms (HAMD-6 and Altman-5), side effects (ASAQ), quality of life (EQ-5D-5L) and work productivity/activity impairment (WPAI).

Safety Patients will follow treatment-as-usual with their clinician being responsible for safety monitoring according to local treatment guidelines. Hence, participation in the present study will not change any aspect of the participants treatment apart that eLi12 potentially can give the clinician additional information on the individual 12-hour Se-Li level.

Sample size At the bipolar outpatient clinic at AUHP, approximately 140 patients are treated with lithium and 80 Se-Li tests are taken each month. At the outpatient clinic for affective disorders at Randers Psychiatric hospital, approximately 180 patients are treated with lithium with 60 Se-Li tests taken each month. At the outpatient clinic for affective disorders at Gødstrup Psychiatric hospital, approximately 50 patients are treated with lithium with 30 Se-Li tests taken each month. The investigators expect that 100, 75, and 25 lithium-treated patients from AUHP, Randers, and Gødstrup will participate in this study, respectively, i.e., 200 in total, with approximately 70 Se-Li tests/month (after full recruitment, which is expected to last 3-6 months at each site). All patients will have to register the time since the last lithium dose at every lithium blood test, independent of randomization status. During the study, patients will be randomized to either 1) have eLi12 shown together with their usual Se-Li measurement or 2) to only have the Se-Li measurement presented (i.e., treatment-as-usual without the eLi12 estimation). Hence, a conservative expectation is >1000 Se-Li blood tests during the study. As for co-primary outcome 1, whether patients are able to register the time of the last lithium dose, the investigators would based on 1000 observations and an expected 80% registering the time for lithium intake correctly be able to get a precision (CI width) of 0.055 with a power of 90%. For the second and third co-primary outcome, based on data from the large proof-of-concept trial, the investigators have 99% power to detect a mean difference of 0.07 between eLi12 and the measured Se-Li concentration.

Study duration Q4 2025 to Q4 2027.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with bipolar disorder (ICD-10: F30-31)
3. Followed at the bipolar disorder outpatient clinic at AUHP, the outpatient clinic for affective disorders at Randers Psychiatric hospital, or the outpatient clinic for affective disorders at Gødstrup Psychiatric hospital
4. Treated with lithium (ATC-code: N05AN01)
5. Able to give informed oral and written consent.

Exclusion Criteria:

1. Any coercive measure in the study period including patients in forensic psychiatry
2. In a clinical condition where the treating clinician evaluates that the patient is not able to attend the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients registering the time since the last lithium dose | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027
The difference between eLi12 and Se-Li | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027
  For each lithium blood test, the difference between the measured Se-Li concentration and the estimated eLi12 level (i.e. for the same blood test based on the patient-reported time since last lithium intake and the Se-Li concentration)
for those periods of time where participants have no change in their lithium dose, the variation in eLi12 compared to the actual measured lithium concentrations at ≤10 hours or ≥14 hours from the last dose | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027

SECONDARY OUTCOMES:
questionnaires filled out before and after participation in the study by the participants whether they prefer a solution as eLi12 that gives more flexibility with regards to timing of lithium blood tests | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027
questionnaires filled out regularly by the attending clinicians reporting whether eLi12 is a safe and intuitive solution | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027
changes on questionnaires filled out by participants before and after the study measuring self-reported symptoms (HAMD-6 and Altman-5), side effects (ASAQ), quality of life (EQ-5D-5L) and work productivity/activity impairment (WPAI). | Each patient participates from the individual randomization date and up to 24 months. Follow-up ends when a participant wants to leave the study or at the end of the study on December 31, 2027

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Clinic for Bipolar Disorder, Aarhus University Hospital Psychiatry, Aarhus
  - Psychiatric Hospital Gødstrup, Herning
  - Psychiatric Hospital Randers, Randers

IPD SHARING:
Plan to Share IPD: No